CLINICAL TRIAL: NCT04941365
Title: Quantifying Systemic Immunosuppression to Personalize Cancer Therapy
Acronym: SERPENTINE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: please refer to NCT05621837
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Fondazione IRCCS ISTITUTO NAZIONALE TUMORI (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROICM 2021-05 SER
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Melanoma; Metastatic Breast Cancer; Advanced Renal Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Non-small Cell Lung Cancer Stage III; Healthy
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This is a multi-centric prospective observational study, testing whether the blood level of MDSC-related immunosuppression does correlate with clinical outcome (clinical response by RECIST criteria, PFS, DFS) and thus may help predicting sensitivity or resistance to therapy in cancer patients. In addition, blood samples will be extensively studied to gain insights into the molecular and metabolic pathways regulating myeloid-mediated immunosuppression, with the goal of defining novel targets of immunomodulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Blood samples will be collected at baseline(Visit 1), and during therapy at visit 2 (around one month after the treatment starting) and at Visit 3 (around three months after the treatment starting. And, optionally, in case of a disease progression (PD).
  Interventions: Diagnostic Test: single arm

INTERVENTIONS:
Diagnostic Test: single arm — Blood samples will be collected at baseline(Visit 1), and during therapy at visit 2 (around one month after the treatment starting) and at Visit 3 (around three months after the treatment starting. And, optionally, in case of a disease progression (PD).

SUMMARY:
It is nowadays well established that the immune system can profoundly influence disease outcome in cancer patients. Increasing evidence is indeed showing that patients displaying spontaneous T cell-mediated immune response against their tumor (defined as immune surveillance) have higher chance to respond to therapies and display globally better prognosis. Conversely, patients whose tumor is characterized by immunosuppression, usually involving myeloid cells and chronic inflammation pathways, often undergo rapid progression and rarely benefit from therapy. Hence, capturing the immune features of individual tumors can help to predict disease course and tailor the therapeutic workup in clinical setting.

DETAILED DESCRIPTION:
It is nowadays well established that the immune system can profoundly influence disease outcome in cancer patients. Increasing evidence is indeed showing that patients displaying spontaneous T cell-mediated immune response against their tumor (defined as immune surveillance) have higher chance to respond to therapies and display globally better prognosis. Conversely, patients whose tumor is characterized by immunosuppression, usually involving myeloid cells and chronic inflammation pathways, often undergo rapid progression and rarely benefit from therapy. Hence, capturing the immune features of individual tumors can help to predict disease course and tailor the therapeutic workup in clinical setting. In addition, overcoming cancer-related immunosuppression could provide a valid tool to rescue immune surveillance and implement cancer treatment through the engagement of the immunological control.

Delivering the right cure to the right patient is the base of precision medicine, and intensive efforts are ongoing worldwide to include the assessment of immune features unto individual patient profiling. However, despite the enormous amount of preclinical and clinical data proving the pivotal role of immunity in molding disease outcome, the immune-related assays that have been introduced into clinical practice, are still scantly. One major limitation is related to the fact that most immune biomarkers have been so far evaluated at tumor site, which implies the need for tumor biopsies and limitations related to intra-lesion heterogeneity. Instead, tests relying on blood samples are easier to perform, more reliable in terms of reproducibility, and repeatable for longitudinal studies. Of note, it is nowadays well established that cancer immunity is a systemic process involving different peripheral immune organs (lymph nodes, bone marrow and spleen) and, as such, it can be measured in blood. Hence, circulating immune cells might represent an informative source of biomarkers to reveal the type and activation status of immunity at single patient level. This holds particularly true for tumor-related immunosuppression, which is mostly mediated myeloid cells and it is responsible for blunting antitumor T cell immune-surveillance. Early during carcinogenesis, cancer cells establish a tight cross-talk with the bone marrow, mediated by tumor-released soluble factors that influence myelopoiesis. This process results in the introduction into the peripheral circulation, of aberrant immunosuppressive myeloid cells, globally known as Myeloid-Derived Suppressor Cells (MDSC). MDSC are among the most potent allies of the tumor cells, whose growth and progression in vivo in favored by MDSC ability to inhibit antitumor T cells, promote angiogenesis and sustain metastatic spread. High numbers of MDSC in blood and tumor site of cancer patients is reproducibly associated with poor prognosis and resistance to therapy, including immunotherapy. Studies in preclinical models have also shown that in vivo removal of MDSC reduces tumor expansion in vivo and confers sensitivity to treatment including immunotherapy, indicating a promising role of these cells as appealing novel therapeutic target in cancer. Unfortunately, the phenotypic and functional features of human MDSC are still poorly understood and need to be extensively investigated in clinical setting.

The members of the SERPENTINE Consortium have substantially contributed to the discovery and the study of MDSC in cancer, acquiring deep knowledge on the phenotypic and functional features of these cells both in human and murine setting. In the present trial? coordinators are committed to translate the predictive/prognostic role of MDSC immune profiling into real-life clinical practice. Through the concerted effort of all Consortium members and the prospective enrolment of blood samples from a comprehensive cancer patients case set, coordinators are going to develop off-the-shelf predictive/prognostic test based on the standardized quantification of MDSC in peripheral blood of cancer patients. In addition, thanks to our multiple expertise, coordinators are going to get deep insights into the biology of human cancer-related MDSC, for the development of novel therapeutic approaches based on rescuing tumor immune surveillance by antagonizing immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of metastatic/locally advanced melanoma, hormone-refractory breast cancer, RCC and UC, SCCHN, SCC or NSCLC, stage III resectable NSCLC will also be included
* Will and ability to comply with the protocol
* Willingness and ability to provide an adequate archival Formalin- Fixed Paraffin-Embedded (FFPE) tumor sample available for exploratory biomarker analysis
* Age from 18 to 90 years at the time of recruitment
* ECOG Performance Status < 2
* Understanding and signature of the informed consent

Exclusion Criteria:

* Known history of HIV infection
* Serious neurological or psychiatric disorders
* Pregnancy or lactation
* Inability or unwillingness of participant to give written informed consent
* Inability or unwillingness to be regularly followed up at the enrolling center

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Investigation of whether a flow cytometry blood-based MDSC quantification assay, does predict disease course in different cancer patients undergoing standard therapies including immunotherapy, chemotherapy, target therapies and surgery. | during 3 months after the start of the treatment
  Correlation of myeloid-related blood biomarkers (including quantification of myeloid cell subsets in peripheral blood mononuclear cells and whole blood) with disease outcome including objective response to therapy, progression-free survival and overall survival, to identify tool for predicting resistance to treatment and poor prognosis.

SECONDARY OUTCOMES:
discovery and development of an additional MDSC-related blood biomarkers associated with the phenotypic or functional profile of these cells | during 3 months after the start of the treatment
  Transcriptional signatures identified on PBMC and sorted myeloid cells form whole blood, at baseline or first evaluation
obtention insights into the signaling and metabolic pathways regulating human MDSC, for the discovery of innovative cancer therapeutic targets based on immunomodulation | during 3 months after the start of the treatment
  Metabolomic profiles, as defined by the concentration of individual metabolites or cluster of metabolites implicated in amino acid and lipid metabolism
perform the first survey assessing the link between MDSC (myeloid-derived suppressor cells) immunosuppression and patient psychological traits, including socio-economical status and perceived social isolation | at the baseline
  Loneliness Questionnaire (no min and max values)
perform the first survey assessing the link between MDSC (myeloid-derived suppressor cells) immunosuppression and patient psychological traits, including socio-economical status and perceived social isolation | at the baseline
  Socio-Economical Questionnaire (no min and max values)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ribas A, Wolchok JD. Cancer immunotherapy using checkpoint blockade. Science. 2018 Mar 23;359(6382):1350-1355. doi: 10.1126/science.aar4060. Epub 2018 Mar 22. PMID 29567705
- [Background] Galluzzi L, Buque A, Kepp O, Zitvogel L, Kroemer G. Immunological Effects of Conventional Chemotherapy and Targeted Anticancer Agents. Cancer Cell. 2015 Dec 14;28(6):690-714. doi: 10.1016/j.ccell.2015.10.012. PMID 26678337
- [Background] Apetoh L, Tesniere A, Ghiringhelli F, Kroemer G, Zitvogel L. Molecular interactions between dying tumor cells and the innate immune system determine the efficacy of conventional anticancer therapies. Cancer Res. 2008 Jun 1;68(11):4026-30. doi: 10.1158/0008-5472.CAN-08-0427. PMID 18519658
- [Background] Peguillet I, Milder M, Louis D, Vincent-Salomon A, Dorval T, Piperno-Neumann S, Scholl SM, Lantz O. High numbers of differentiated effector CD4 T cells are found in patients with cancer and correlate with clinical response after neoadjuvant therapy of breast cancer. Cancer Res. 2014 Apr 15;74(8):2204-16. doi: 10.1158/0008-5472.CAN-13-2269. Epub 2014 Feb 17. PMID 24535711
- [Background] Wilmott JS, Long GV, Howle JR, Haydu LE, Sharma RN, Thompson JF, Kefford RF, Hersey P, Scolyer RA. Selective BRAF inhibitors induce marked T-cell infiltration into human metastatic melanoma. Clin Cancer Res. 2012 Mar 1;18(5):1386-94. doi: 10.1158/1078-0432.CCR-11-2479. Epub 2011 Dec 12. PMID 22156613
- [Background] Thorsson V, Gibbs DL, Brown SD, Wolf D, Bortone DS, Ou Yang TH, Porta-Pardo E, Gao GF, Plaisier CL, Eddy JA, Ziv E, Culhane AC, Paull EO, Sivakumar IKA, Gentles AJ, Malhotra R, Farshidfar F, Colaprico A, Parker JS, Mose LE, Vo NS, Liu J, Liu Y, Rader J, Dhankani V, Reynolds SM, Bowlby R, Califano A, Cherniack AD, Anastassiou D, Bedognetti D, Mokrab Y, Newman AM, Rao A, Chen K, Krasnitz A, Hu H, Malta TM, Noushmehr H, Pedamallu CS, Bullman S, Ojesina AI, Lamb A, Zhou W, Shen H, Choueiri TK, Weinstein JN, Guinney J, Saltz J, Holt RA, Rabkin CS; Cancer Genome Atlas Research Network; Lazar AJ, Serody JS, Demicco EG, Disis ML, Vincent BG, Shmulevich I. The Immune Landscape of Cancer. Immunity. 2018 Apr 17;48(4):812-830.e14. doi: 10.1016/j.immuni.2018.03.023. Epub 2018 Apr 5. PMID 29628290
- [Background] Spitzer MH, Carmi Y, Reticker-Flynn NE, Kwek SS, Madhireddy D, Martins MM, Gherardini PF, Prestwood TR, Chabon J, Bendall SC, Fong L, Nolan GP, Engleman EG. Systemic Immunity Is Required for Effective Cancer Immunotherapy. Cell. 2017 Jan 26;168(3):487-502.e15. doi: 10.1016/j.cell.2016.12.022. Epub 2017 Jan 19. PMID 28111070
- [Background] Dumeaux V, Fjukstad B, Fjosne HE, Frantzen JO, Holmen MM, Rodegerdts E, Schlichting E, Borresen-Dale AL, Bongo LA, Lund E, Hallett M. Interactions between the tumor and the blood systemic response of breast cancer patients. PLoS Comput Biol. 2017 Sep 28;13(9):e1005680. doi: 10.1371/journal.pcbi.1005680. eCollection 2017 Sep. PMID 28957325
- [Background] Cortez-Retamozo V, Etzrodt M, Newton A, Rauch PJ, Chudnovskiy A, Berger C, Ryan RJ, Iwamoto Y, Marinelli B, Gorbatov R, Forghani R, Novobrantseva TI, Koteliansky V, Figueiredo JL, Chen JW, Anderson DG, Nahrendorf M, Swirski FK, Weissleder R, Pittet MJ. Origins of tumor-associated macrophages and neutrophils. Proc Natl Acad Sci U S A. 2012 Feb 14;109(7):2491-6. doi: 10.1073/pnas.1113744109. Epub 2012 Jan 30. PMID 22308361
- [Background] Gabrilovich DI. Myeloid-Derived Suppressor Cells. Cancer Immunol Res. 2017 Jan;5(1):3-8. doi: 10.1158/2326-6066.CIR-16-0297. PMID 28052991
- [Background] Groth C, Hu X, Weber R, Fleming V, Altevogt P, Utikal J, Umansky V. Immunosuppression mediated by myeloid-derived suppressor cells (MDSCs) during tumour progression. Br J Cancer. 2019 Jan;120(1):16-25. doi: 10.1038/s41416-018-0333-1. Epub 2018 Nov 9. PMID 30413826
- [Background] Ostrand-Rosenberg S. Myeloid derived-suppressor cells: their role in cancer and obesity. Curr Opin Immunol. 2018 Apr;51:68-75. doi: 10.1016/j.coi.2018.03.007. Epub 2018 Mar 13. PMID 29544121
- [Background] Wesolowski R, Markowitz J, Carson WE 3rd. Myeloid derived suppressor cells - a new therapeutic target in the treatment of cancer. J Immunother Cancer. 2013 Jul 15;1:10. doi: 10.1186/2051-1426-1-10. eCollection 2013. PMID 24829747
- [Background] Fleming V, Hu X, Weber R, Nagibin V, Groth C, Altevogt P, Utikal J, Umansky V. Targeting Myeloid-Derived Suppressor Cells to Bypass Tumor-Induced Immunosuppression. Front Immunol. 2018 Mar 2;9:398. doi: 10.3389/fimmu.2018.00398. eCollection 2018. PMID 29552012
- [Background] Engblom C, Pfirschke C, Pittet MJ. The role of myeloid cells in cancer therapies. Nat Rev Cancer. 2016 Jul;16(7):447-62. doi: 10.1038/nrc.2016.54. PMID 27339708
- [Background] Filipazzi P, Valenti R, Huber V, Pilla L, Canese P, Iero M, Castelli C, Mariani L, Parmiani G, Rivoltini L. Identification of a new subset of myeloid suppressor cells in peripheral blood of melanoma patients with modulation by a granulocyte-macrophage colony-stimulation factor-based antitumor vaccine. J Clin Oncol. 2007 Jun 20;25(18):2546-53. doi: 10.1200/JCO.2006.08.5829. PMID 17577033
- [Background] Filipazzi P, Huber V, Rivoltini L. Phenotype, function and clinical implications of myeloid-derived suppressor cells in cancer patients. Cancer Immunol Immunother. 2012 Feb;61(2):255-263. doi: 10.1007/s00262-011-1161-9. Epub 2011 Nov 27. PMID 22120756
- [Background] Blattner C, Fleming V, Weber R, Himmelhan B, Altevogt P, Gebhardt C, Schulze TJ, Razon H, Hawila E, Wildbaum G, Utikal J, Karin N, Umansky V. CCR5+ Myeloid-Derived Suppressor Cells Are Enriched and Activated in Melanoma Lesions. Cancer Res. 2018 Jan 1;78(1):157-167. doi: 10.1158/0008-5472.CAN-17-0348. Epub 2017 Oct 31. PMID 29089297
- [Background] Huber V, Vallacchi V, Fleming V, Hu X, Cova A, Dugo M, Shahaj E, Sulsenti R, Vergani E, Filipazzi P, De Laurentiis A, Lalli L, Di Guardo L, Patuzzo R, Vergani B, Casiraghi E, Cossa M, Gualeni A, Bollati V, Arienti F, De Braud F, Mariani L, Villa A, Altevogt P, Umansky V, Rodolfo M, Rivoltini L. Tumor-derived microRNAs induce myeloid suppressor cells and predict immunotherapy resistance in melanoma. J Clin Invest. 2018 Dec 3;128(12):5505-5516. doi: 10.1172/JCI98060. Epub 2018 Nov 5. PMID 30260323
- [Background] Bronte V, Brandau S, Chen SH, Colombo MP, Frey AB, Greten TF, Mandruzzato S, Murray PJ, Ochoa A, Ostrand-Rosenberg S, Rodriguez PC, Sica A, Umansky V, Vonderheide RH, Gabrilovich DI. Recommendations for myeloid-derived suppressor cell nomenclature and characterization standards. Nat Commun. 2016 Jul 6;7:12150. doi: 10.1038/ncomms12150. PMID 27381735
- [Background] De Henau O, Rausch M, Winkler D, Campesato LF, Liu C, Cymerman DH, Budhu S, Ghosh A, Pink M, Tchaicha J, Douglas M, Tibbitts T, Sharma S, Proctor J, Kosmider N, White K, Stern H, Soglia J, Adams J, Palombella VJ, McGovern K, Kutok JL, Wolchok JD, Merghoub T. Overcoming resistance to checkpoint blockade therapy by targeting PI3Kgamma in myeloid cells. Nature. 2016 Nov 17;539(7629):443-447. doi: 10.1038/nature20554. Epub 2016 Nov 9. PMID 27828943
- [Background] Welters MJ, van der Sluis TC, van Meir H, Loof NM, van Ham VJ, van Duikeren S, Santegoets SJ, Arens R, de Kam ML, Cohen AF, van Poelgeest MI, Kenter GG, Kroep JR, Burggraaf J, Melief CJ, van der Burg SH. Vaccination during myeloid cell depletion by cancer chemotherapy fosters robust T cell responses. Sci Transl Med. 2016 Apr 13;8(334):334ra52. doi: 10.1126/scitranslmed.aad8307. PMID 27075626
- [Background] Crunkhorn S. Cancer: New path to improving immunotherapy. Nat Rev Drug Discov. 2018 Mar;17(3):164. doi: 10.1038/nrd.2018.22. Epub 2018 Feb 16. No abstract available. PMID 29449711